CLINICAL TRIAL: NCT03863951
Title: The Study on the Association of Intestinal Flora and Early Post-stroke Depression in Patients With Acute Ischemic Stroke
Brief Title: Poststroke Depression of Clinical Trial Registration
Acronym: IFEPSDAIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2018-024
Record Dates: First submitted 2019-02-24; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-01

CONDITIONS: Stroke; Depression
Keywords: ischemic stroke; depression; intestinal microbiota
MeSH Terms: conditions — Stroke; Depression; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with poststroke depression: No intervention
- Patients without poststroke depression: No intervention

SUMMARY:
The investigators aim to explore the relationship between gut microbiota composition and earlier poststroke depression via 16S rRNA sequencing.

DETAILED DESCRIPTION:
In this study, patients with first ever acute ischemic stroke were studied. According to the psychological assessment, patients were divided into two groups according to whether or not there was a PSD at the earlier stage of stroke. Clinical biological data and blood and feces samples were collected. Firstly, 16srDNA sequencing was used to study the difference in the composition and diversity of intestinal microbial communities in the two groups of patients. Then the two groups selected individual representative samples and conducted macro genome sequencing. At the same time, by analyzing the correlation between the intestinal flora and the clinical risk factors and neurotransmitters in early PSD patients, the key functional bacteria related to PSD were identified.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with the first ever acute ischemic stroke occurring within 2 weeks and were confirmed by CT or MRI,
* has no history of depression or use of antidepressants or antipsychotics,
* were competent to consent to take part in this research.

Exclusion Criteria:

* significant acute or severe illness such as infection,heart failure and tumor,
* previous diagnosis of depression or other mental disorder or who had recently accepted antidepressants or antipsychotics,
* antibiotics in the last two weeks,
* severe aphasia or dysarthria,irritable bowel syndrome,asthma,and pregnant or lactating women,
* a previous history of neurological illness including AD and PD，
* Inflammatory bowel disease，

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The Composition of Intestinal Microbial Communities Calculated by OTU Analysis | 2 weeks
  The composition were measured in number based on OTU data
The Diversity of Intestinal Microbial Communities Calculated by OTU Analysis | 2 weeks
  Community diversity measured in the Shannon index
The Poststroke Depression Assessed by Hamilton Rating Scale for Depression (HAMD-17) Score | 3 months
  Mild depression（HAMD-17 Score>7，≤17）, moderate depression（HAMD-17 Score>17，≤24）, major depression（HAMD-17 Score>24）
Functional Independence Assessed by Modified Rankin Scale (mRS）score | 3 months
  MRS score range from 0 to 6. Favourable outcome (mRS score≤2), worse outcome (mRS score>2), and death (mRS score = 6).

SECONDARY OUTCOMES:
The Plasma Level of 5-Hydroxytryptamine( 5-HT) Neurotransmitter Using Enzyme-Linked Immunosorbent Assay ( ELISA) Methods | 2 weeks
  5-HT measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Yurong Zhang, PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Yurong Zhang, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No